CLINICAL TRIAL: NCT07168304
Title: Clinical Outcome of Zinc Plus Saccharomyces Boulardii Versus Zinc Alone in the Treatment of Acute Diarrhea in Children Under 5 Years of Age
Brief Title: Zinc Plus Saccharomyces Boulardii Versus Zinc Alone in the Treatment of Acute Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Hammad-Multan
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Watery Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Standard treatment plus S. boulardii
  Interventions: Drug: S. boulardii
- No probiotic group (No Intervention): Standard treatment only

INTERVENTIONS:
Drug: S. boulardii — Participants received zinc plus S. boulardii supplementation according to the World Health Organization recommendations.
  Arms: Probiotic group

SUMMARY:
In literature combined therapy of zinc with S. boulardii in the treatment of acute diarrhea has not been addressed satisfactorily in the recent past. Therefore, this study was planned aiming to compare the mean time taken to resolve diarrhea and the mean time taken to resolve vomiting in children under 5 years of age having acute diarrhea with zinc plus S. boulardii versus zinc alone.

DETAILED DESCRIPTION:
Zinc has been used as a recommended choice treating acute watery ailments among children. If any significant beneficial effect in the combined efficacy of zinc with S. boulardii is found, it may add on to pre-existing knowledge and may lead clinicians to delineate the treatment guidelines to provide more effective treatment to the patients in clinical practices to reduce undesirable morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender
* Aged between 1 month up to 5 years
* Presented with acute diarrhea

Exclusion Criteria:

* Children with concurrent acute illnesses (meningitis, sepsis, or pneumonia)
* Severe chronic conditions (cystic fibrosis, endocrinopathies, food allergies, or chronic gastrointestinal diseases)
* Severe undernutrition (weight-for-age <60% of the 50th percentile of CDC 2000 standards)
* Children who used probiotics, antibiotics, or anti-diarrheal drugs within the past 7 days
* The presence of visible blood in stools

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhea | 7 days
  The duration from initiation of treatment until passage of normal stools (Bristol Stool Form Scale types 3-4).
Resolution of vomiting | 14 hours
  The time from the start of treatment to the last episode of vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hammad Riaz, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan
Locations (1):
- The Children's Hospital and The Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.